CLINICAL TRIAL: NCT01443130
Title: A Randomized, Controlled Clinical Trial of Chloroquine as Chemoprophylaxis Versus Intermittent Preventive Therapy to Prevent Malaria in Pregnancy in Malawi
Brief Title: Chloroquine for Malaria in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0112; 4R01AI104702-04 (NIH)
Record Dates: First submitted 2011-09-01; First posted 2011-09-29 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2015-05

CONDITIONS: Malaria
Keywords: malaria,Malawi,pregnancy
MeSH Terms: conditions — Malaria | interventions — Chloroquine; fanasil, pyrimethamine drug combination

ARMS (3):
- Chloroquine IPT (Experimental): 300 subjects to receive a therapeutic dose of chloroquine (1,500 mg given over 3 days, 2 tablets on Day 0, 2 tablets on Day 1, 1 tablet on Day 2) will be administered twice during pregnancy at 20-28 weeks and at 28-34 weeks.
  Interventions: Drug: Chloroquine
- Chloroquine Prophylaxis (Experimental): 300 subjects to receive a loading dose of chloroquine (base) 600 mg (2 tablets) at first administration followed by 300 mg of chloroquine base (1 tablet) every week.
  Interventions: Drug: Chloroquine
- SP IPT (Active Comparator): 300 subjects to receive a therapeutic dose of sulfadoxine-pyrimethamine (SP), (1500 mg sulfadoxine and 75 mg pyrimethamine (3 tablets)) administered twice during pregnancy at 20-28 weeks and at 28-34 weeks.
  Interventions: Drug: Sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Chloroquine — Chloroquine tablets contain 300 mg chloroquine base per tablet. Dosages: Chloroquine 1,500 mg base over 3 days twice during pregnancy or Chloroquine 600 mg loading dose followed by 300 mg orally once per week. Intermittant preventative treatment in pregnancy (IPTp) doses will be administered between weeks 20-28 and weeks 28-34 gestation, 4 weeks apart. Participants randomized to IPTp with chloroquine will require their second and third doses of chloroquine after the initial dose given in the clinic and those assigned to chloroquine chemoprophylaxis will require weekly doses.
  Arms: Chloroquine IPT; Chloroquine Prophylaxis
Drug: Sulfadoxine-pyrimethamine — Sulfadoxine-pyrimethamine 3 tablets (1,500 mg sulfadoxine and 75 mg pyrimethamine) twice during pregnancy. Intermittant preventive treatment in pregnancy (IPTp) doses will be administered between weeks 20-28 and weeks 28-34, 4 weeks apart.
  Arms: SP IPT

SUMMARY:
The purpose of this study is to test prevention strategies for pregnancy-related malaria. Researchers will compare different malaria treatments and treatment schedules which include chloroquine therapy (weekly doses versus being dosed twice during pregnancy for 3 days each time) to the standard practice of preventive treatment intervals in pregnancy (with the drug sulfadoxine-pyrimethamine given twice during pregnancy). Participants will include 900 pregnant women, who will be assigned to one of three treatment groups. Blood samples will be collected at every visit before birth and any time the participant is ill to determine if malaria is present. Pregnant women will be monitored during pregnancy and newborns will be assessed at birth and followed until about 14 weeks. Participant involvement in the study is expected to last about 12 months.

DETAILED DESCRIPTION:
In areas of high malaria endemicity, typical of much of sub-Saharan Africa, despite having achieved semi-immunity to malaria in adulthood, women become vulnerable to malaria infection during pregnancy, especially during their first or second pregnancy. They have increased rates of infection in the peripheral blood and high concentrations of parasites can be found in the placenta. On histological examination, mature asexual parasites, forms that are not usually detected in the peripheral blood, accumulate in the placenta. Pregnancy-specific variant surface antigens are responsible for the increased vulnerability of pregnant women to malaria because they are unrecognized by the immune systems of women who encounter them for the first time in their first pregnancy. In subsequent pregnancies, women develop immunity to these parasite surface antigens and the parasites are cleared by the host response. Plasmodium (P) falciparum infection during pregnancy has important health consequences for both pregnant women and their newborns. Adverse outcomes of pregnancy-associated malaria that have been documented in Malawi include maternal anemia, low birth weight (LBW), and increased infant mortality. The primary objective of the study is to compare weekly chloroquine prophylaxis and chloroquine intermittent preventative therapy (IPT) for malaria in pregnancy (IPTp) to the standard practice [IPTp with sulfadoxine-pyrimethamine (SP)] with respect to prevention of placental malaria. The secondary objectives are: to compare weekly chloroquine prophylaxis and chloroquine IPTp to the standard practice (IPTp with SP) with respect to prevention of malaria during pregnancy; to compare weekly chloroquine prophylaxis and chloroquine IPTp to the standard practice (IPTp with SP) with respect to prevention of the adverse maternal and newborn effects of pregnancy-associated malaria. The exploratory objective identify the vulnerable periods during pregnancy when malaria infection is more likely to cause placental infection, maternal anemia, and low infant birth weight. This is a randomized controlled trial to compare chloroquine as IPT or chloroquine as chemoprophylaxis to IPTp with SP. Women will be randomized after Screening and enrollment, and they begin the assigned treatment between Week 20 and Week 28 gestation. Specimens will be collected at every prenatal visit and any time the participant is ill to determine if malaria is present. Pregnant women will be monitored during pregnancy, and newborns will be assessed at birth and followed until they are approximately 14 weeks of age. Participants will be randomized to one of the following regimens: Chloroquine approximately 1,500 mg base over 3 days, twice during pregnancy (2 tablets on Day 0, 2 tablets on Day 1, 1 tablet on Day 2); Chloroquine base 600 mg (2 tablets) loading dose followed by 300 mg (1 tablet) orally once per week until delivery; SP 1500 mg/75 mg twice during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Women who present to the Ndirande Antenatal Clinic (ANC) and meet the following inclusion criteria will be enrolled in the study: -Before the end of 27th week of gestation -First or second pregnancy -Anticipate remaining in Blantyre until 14 weeks after delivery -Agree to deliver at the Ndirande Health Centre or Queen Elizabeth Central Hospital (QECH) -Provision of informed consent

Exclusion Criteria:

-Chronic use (>14 days) of any medication with antimalarial or antifolate activity -Human immunodeficiency virus (HIV) infection -Known high-risk pregnancy requiring regular supervision of an obstetrician -Allergy to any of the study drugs

Max Age: 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Blantyre Malaria Project - Queen Elizabeth Central Hospital, Blantryre, Blantyre, Malawi

REFERENCES:
- [Derived] Buchwald AG, Boudova S, Peterson I, Divala T, Mungwira R, Mawindo P, Gladstone M, Cairo C, Laufer MK. The Association among Malaria in Pregnancy, Neonatal inflammation, and Neurocognitive Development in a Cohort of Malawian Infants. Am J Trop Med Hyg. 2022 Oct 17;107(5):1036-1040. doi: 10.4269/ajtmh.22-0409. Print 2022 Nov 14. PMID 36252805
- [Derived] Patson N, Mukaka M, Kazembe L, Eijkemans MJC, Mathanga D, Laufer MK, Chirwa T. Comparison of statistical methods for the analysis of recurrent adverse events in the presence of non-proportional hazards and unobserved heterogeneity: a simulation study. BMC Med Res Methodol. 2022 Jan 20;22(1):24. doi: 10.1186/s12874-021-01475-8. PMID 35057743
- [Derived] Patson N, Mukaka M, Peterson I, Divala T, Kazembe L, Mathanga D, Laufer MK, Chirwa T. Effect of adverse events on non-adherence and study non-completion in malaria chemoprevention during pregnancy trial: A nested case control study. PLoS One. 2022 Jan 19;17(1):e0262797. doi: 10.1371/journal.pone.0262797. eCollection 2022. PMID 35045119
- [Derived] Divala TH, Mungwira RG, Mawindo PM, Nyirenda OM, Kanjala M, Ndaferankhande M, Tsirizani LE, Masonga R, Muwalo F, Boudova S, Potter GE, Kennedy J, Goswami J, Wylie BJ, Muehlenbachs A, Ndovie L, Mvula P, Mbilizi Y, Tomoka T, Laufer MK. Chloroquine as weekly chemoprophylaxis or intermittent treatment to prevent malaria in pregnancy in Malawi: a randomised controlled trial. Lancet Infect Dis. 2018 Oct;18(10):1097-1107. doi: 10.1016/S1473-3099(18)30415-8. Epub 2018 Sep 5. PMID 30195996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were pregnant women in their first or second pregnancy recruited during presentation at the Ndirande Antenatal Clinic (ANC) at the Ndirande Health Centre, enrolled between 22 February 2012 and 16 May 2014.
Pre-assignment Details: The infants born to these participants were also enrolled in the study to be assessed at birth and followed to 14 weeks. The infants are reported here as separate arms of the study, grouped by the study product given to the mother.
Groups:
- Maternal Chloroquine Prophylaxis: Maternal participants receive a loading dose of chloroquine (base) 600 mg (2 tablets) at first administration followed by 300 mg of chloroquine base (1 tablet) every week until delivery.
- Maternal Chloroquine IPT: Maternal participants receive a therapeutic dose of chloroquine (1,500 mg given over 3 days, 2 tablets on Day 0, 2 tablets on Day 1, 1 tablet on Day 2) administered twice during pregnancy at 20-28 weeks and at 28-34 weeks.
- Maternal SP IPT: Maternal participants receive a therapeutic dose of sulfadoxine-pyrimethamine (SP), (1500 mg sulfadoxine and 75 mg pyrimethamine (3 tablets)) administered twice during pregnancy at 20-28 weeks and at 28-34 weeks.
- Infant Chloroquine Prophylaxis: Infants born to maternal participants who received chloroquine prophylaxis.
- Infant Chloroquine IPT: Infants born to maternal participants who received chloroquine IPT.
- Infant SP IPT: Infants born to maternal participants who received SP IPT.
Period: Overall Study
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT
Started | 300 | 300 | 300 | 270 | 274 | 259
Completed | 232 | 231 | 223 | 231 | 230 | 225
Not Completed | 68 | 69 | 77 | 39 | 44 | 34
Not completed — Lost to Follow-up | 44 | 42 | 50 | 23 | 25 | 21
Not completed — Death | 0 | 1 | 0 | 7 | 10 | 8
Not completed — Adverse Event | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 3 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 15 | 14 | 12 | 7 | 7 | 2
Not completed — Death of Subject's Infant | 5 | 10 | 11 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study are included in the baseline analysis population, with the exception of the age continuous for all groups, which is limited to the maternal participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT | Total
Number analyzed (Participants) | 300 | 300 | 300 | 270 | 274 | 259 | 1703
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 99 | 81 | 90 | 270 | 274 | 259 | 1073
  Between 18 and 65 years | 201 | 219 | 210 | 0 | 0 | 0 | 630
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.40 (3.59) | 20.67 (3.24) | 20.44 (3.14) | 0 (0) | 0 (0) | 0 (0) | 20.50 (3.33)
Gender [Count of Participants; unit: Participants]
  Female | 300 | 300 | 300 | 133 | 143 | 136 | 1312
  Male | 0 | 0 | 0 | 137 | 131 | 123 | 391
Region of Enrollment [Number; unit: participants]
  Malawi | 300 | 300 | 300 | 270 | 274 | 259 | 1703

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Placental Malaria Infection Based on Histology
Description: The placenta was collected at the time of delivery for examination by histology to determine malaria infection. Malaria infection was concluded if histology identified parasites or malaria pigment in the placental tissue.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: All participants from whom the placental histopathology slides collected at the time of delivery were reviewed are included in the analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of pregnancies
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 259 | 253 | 253
percentage of pregnancies | 11.58 [7.52 to 16.80] | 15.42 [10.67 to 21.21] | 15.42 [10.67 to 21.21]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of placental malaria infection based on histology is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.2441, Fisher Exact — A Bonferroni correction was used due to multiple comparisons. Comparisons are statistically significant if the two-sided p-value is ≤ 0.05/2=0.025
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of placental malaria infection based on histology is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Incidence of Placental Malaria by Placental Impression Smear
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of malaria infection in the placenta based on diagnosis by positive placental impression smear results.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all maternal participants whose pregnancies were followed to delivery and from whom a placenta was collected and an impression smear performed.
Measure: Number (97.5% Confidence Interval); unit: percentage of placentas
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 259 | 254 | 253
percentage of placentas | 0 [0.00 to 1.68] | 0 [0.00 to 1.71] | 0.40 [0.00 to 2.50]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of malaria by placental impression smear is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4941, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of malaria by placental impression smear is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4990, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Incidence of Maternal Anemia (Hemoglobin < 10 Grams/Deciliter)
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of anemia among maternal participants during pregnancy . Anemia is defined as having a hemoglobin value less than 10 grams/deciliter (gm/dL).
Time Frame: From enrollment until delivery, approximately 12-36 weeks
Population: The analysis population includes all maternal participants.
Measure: Number (97.5% Confidence Interval); unit: percentage of maternal participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 300 | 300 | 300
percentage of maternal participants | 18.3 [13.58 to 23.89] | 23.7 [18.36 to 29.64] | 22.0 [16.85 to 27.86]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of maternal anemia is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.3089, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of maternal anemia is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.6973, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Incidence of Maternal Severe Anemia (Hemoglobin < 7gm/dl)
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of severe anemia among maternal participants during pregnancy. Severe anemia is defined as having a hemoglobin value less than 7 gm/dl.
Time Frame: From enrollment until delivery, approximately 12-36 weeks
Population: The analysis population includes all maternal participants.
Measure: Number (97.5% Confidence Interval); unit: percentage of maternal participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 300 | 300 | 300
percentage of maternal participants | 0.0 [0.00 to 1.45] | 0.3 [0.00 to 2.11] | 0.3 [0.00 to 2.11]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of maternal severe anemia is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of maternal severe anemia is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Incidence of Stillbirth
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of participants' deliveries whose outcome was stillbirth, defined as an infant born without any signs of life at 28 weeks or greater of gestation.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all participants whose pregnancies were followed to delivery.
Measure: Number (97.5% Confidence Interval); unit: percentage of deliveries
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 272 | 273 | 263
percentage of deliveries | 1.10 [0.17 to 3.54] | 0.37 [0.00 to 2.31] | 1.90 [0.52 to 4.78]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of stillbirth is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4979, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of stillbirth is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.1166, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Incidence of Miscarriage
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of participants' deliveries whose outcome was miscarriage, defined as an infant delivered without any signs of life at less than 28 weeks of gestation.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all maternal participants.
Measure: Number (97.5% Confidence Interval); unit: percentage of pregnancies
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 300 | 300 | 300
percentage of pregnancies | 0.33 [0 to 2.11] | 0.67 [0.06 to 2.68] | 1.00 [0.16 to 3.21]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of miscarriage is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.6237, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of miscarriage is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Incidence of Preterm Delivery
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of participants' deliveries whose outcome was preterm delivery, defined as delivery less than 37 weeks of gestation. The outcome of the delivery was not considered, and could have been live birth, stillbirth, or miscarriage.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all participants whose pregnancies were followed to delivery.
Measure: Number (97.5% Confidence Interval); unit: percentage of deliveries
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 272 | 273 | 263
percentage of deliveries | 8.46 [5.08 to 13.02] | 9.89 [6.23 to 14.69] | 6.84 [3.80 to 11.17]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of preterm delivery is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.5187, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of preterm delivery is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.2163, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Infant Mortality Rate to 14 Weeks of Age
Description: Infants were followed from the time of delivery until 14 weeks of age. This outcome measure provides the incidence of infants who died within 14 weeks of delivery.
Time Frame: For 14 weeks after delivery.
Population: The analysis population includes all enrolled infants.
Measure: Number (97.5% Confidence Interval); unit: percentage of infants
Arm/Group | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT
Number analyzed (Participants) | 270 | 274 | 259
percentage of infants | 2.22 [0.70 to 5.18] | 3.65 [1.58 to 7.07] | 3.09 [1.18 to 6.46]
Statistical Analysis 1: Comparison: Infant Chloroquine Prophylaxis vs Infant SP IPT; The null hypothesis is the incidence of infant mortality within 14 weeks of delivery is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.5959, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Infant Chloroquine IPT vs Infant SP IPT; The null hypothesis is the incidence of infant mortality within 14 weeks of delivery is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.8127, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Incidence of Low Birth Weight (LBW) (Birthweight < 2500 Grams)
Description: Maternal participants were followed to outcome of the pregnancy. The outcome measure provides the incidence of infants whose birthweight was less than 2500 grams.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all infants born alive with weight data collected at birth.
Measure: Number (97.5% Confidence Interval); unit: percentage of infants
Arm/Group | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT
Number analyzed (Participants) | 263 | 264 | 256
percentage of infants | 15.59 [10.91 to 21.28] | 10.98 [7.06 to 16.05] | 12.11 [7.93 to 17.44]
Statistical Analysis 1: Comparison: Infant Chloroquine Prophylaxis vs Infant SP IPT; The null hypothesis is the incidence of low birth weight is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.2566, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Infant Chloroquine IPT vs Infant SP IPT; The null hypothesis is the incidence of low birth weight is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.7839, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Incidence of Intrauterine Growth Restriction (IUGR)
Description: Infants were followed from the time of delivery until 14 weeks of age. This outcome measure provides the incidence of infants with IUGR at delivery. IUGR is defined as weight below the 10th percentile for gestational age based on the World Health Organization (WHO) fetal growth curve. This classification is supported by literature resulting from the INTERGROWTH-21st Project; José Villar.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: This analysis population includes all infants with weight captured at delivery and with mothers having reported gestational age at delivery.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT
Number analyzed (Participants) | 260 | 261 | 250
percentage of participants | 16.54 [11.70 to 22.37] | 18.01 [12.98 to 23.98] | 20.80 [15.32 to 27.17]
Statistical Analysis 1: Comparison: Infant Chloroquine Prophylaxis vs Infant SP IPT; The null hypothesis is the incidence of intrauterine growth restriction is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.2553, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Infant Chloroquine IPT vs Infant SP IPT; The null hypothesis is the incidence of intrauterine growth restriction is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4354, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Incidence of Active Placental Malaria Infection
Description: Maternal participants were followed to outcome of the pregnancy. This outcome measure provides the number of placental malaria infections in maternal subjects diagnosed by the presence of parasites and/or pigment on histological section or molecular evidence of infection (PCR).
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: This analysis population includes all maternal subjects with placental slides reviewed and PCR results obtained.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 259 | 253 | 253
percentage of participants | 3.09 [1.18 to 6.46] | 3.16 [1.21 to 6.61] | 4.74 [2.24 to 8.67]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of active placental malaria infection is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.3690, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of active placental malaria infection is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4947, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Incidence of Malaria Infection, All Species.
Description: Maternal participants were followed to outcome of the pregnancy. This outcome measure provides the number of malaria infection episodes measured by positive parasitemia in maternal subjects.
Time Frame: Enrollment to delivery (approximately 12-36 weeks)
Population: The analysis population includes all maternal participants.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants | 0.67 [0.06 to 2.68] | 1.67 [0.45 to 4.20] | 3.00 [1.22 to 6.03]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of malaria infection (all species) measured by positive parasitemia is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.0630, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of malaria infection (all species) measured by positive parasitemia is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4184, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Incidence of Clinical Malaria, All Species
Description: Maternal participants were followed to outcome of the pregnancy. Clinical malaria is defined as malaria infection at any parasite density with associated symptoms including at least one of the following: objective fever measured at the clinic, history of fever in the past 48 hours or other symptoms in the last 48 hours including: headache, myalgia, vomiting, or weakness.
Time Frame: Enrollment to delivery (approximately 12-36 weeks)
Population: The analysis population includes all maternal participants.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants | 0.67 [0.53 to 4.89] | 1.33 [0.97 to 6.09] | 3.00 [0.07 to 3.20]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of clinical malaria (all species) is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.0268, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of clinical malaria (all species) is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.1646, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Incidence of Infection in the Fetal Circulation
Description: Maternal participants were followed to outcome of the pregnancy. This outcome measure provides the number of positive for malaria cord blood smear and cord PCR results in maternal subjects based on the results of the thick smear and PCR from the cord blood sample.
Time Frame: At delivery: Approximately 12-36 weeks after enrollment
Population: The analysis population includes all maternal participants with cord blood smears and cord PCR results obtained.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT
Number analyzed (Participants) | 257 | 252 | 251
percentage of participants | 1.95 [0.53 to 4.89] | 2.78 [0.97 to 6.09] | 0.80 [0.07 to 3.20]
Statistical Analysis 1: Comparison: Maternal Chloroquine Prophylaxis vs Maternal SP IPT; The null hypothesis is the incidence of infection in the fetal circulation is identical between subjects receiving maternal chloroquine prophylaxis vs. maternal SP IPT; Test type: Superiority or Other; p = 0.4501, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maternal Chloroquine IPT vs Maternal SP IPT; The null hypothesis is the incidence of infection in the fetal circulation is identical between subjects receiving maternal chloroquine IPT vs. maternal SP IPT; Test type: Superiority or Other; p = 0.1758, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected after the administration of the first dose of study drug throughout the duration of the follow-up period (approximately 14 weeks following delivery).
Arm/Group | Maternal Chloroquine Prophylaxis | Maternal Chloroquine IPT | Maternal SP IPT | Infant Chloroquine Prophylaxis | Infant Chloroquine IPT | Infant SP IPT
Serious Adverse Events (participants affected / at risk) | 23/300 | 29/300 | 26/300 | 46/270 | 65/274 | 43/259
Other Adverse Events (participants affected / at risk) | 255/300 | 251/300 | 234/300 | 195/270 | 186/274 | 171/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Chloroquine Prophylaxis (N=300) | Maternal Chloroquine IPT (N=300) | Maternal SP IPT (N=300) | Infant Chloroquine Prophylaxis (N=270) | Infant Chloroquine IPT (N=274) | Infant SP IPT (N=259)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brief psychotic disorder, with postpartum onset (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accessory auricle (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (9) | 6 (6)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Umbilical cord haemorrhage (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death neonatal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 1 (1)
Group B streptococcus neonatal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 10 (10) | 12 (12)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 9 (9) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 8 (8)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Melanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vacuum extractor delivery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Chloroquine Prophylaxis (N=300) | Maternal Chloroquine IPT (N=300) | Maternal SP IPT (N=300) | Infant Chloroquine Prophylaxis (N=270) | Infant Chloroquine IPT (N=274) | Infant SP IPT (N=259)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 20 (21) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 16 (16) | 19 (21) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 78 (92) | 73 (90) | 62 (77) | 4 (4) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 36 (39) | 28 (29) | 16 (17) | 9 (9) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 17 (20) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 32 (37) | 63 (75) | 16 (17) | 3 (3) | 6 (6) | 4 (4)
Pain (General disorders) | 16 (18) | 26 (30) | 21 (21) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 20 (23) | 10 (12) | 18 (19) | 9 (10) | 9 (9) | 3 (3)
Tonsillitis (Infections and infestations) | 23 (25) | 12 (13) | 12 (15) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 90 (113) | 65 (70) | 73 (82) | 136 (172) | 124 (154) | 118 (152)
Urinary tract infection (Infections and infestations) | 25 (29) | 27 (28) | 27 (28) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 11 (13) | 17 (18) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 12 (12) | 12 (12) | 20 (20) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (25) | 19 (21) | 16 (16) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 79 (88) | 75 (95) | 56 (70) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 16 (16) | 62 (75) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 88 (113) | 76 (96) | 76 (89) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 24 (24) | 28 (28) | 26 (27) | 0 (0) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 20 (20) | 25 (25) | 22 (22) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (11) | 24 (24) | 15 (15) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 12 (15) | 20 (24) | 12 (16) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1) | 7 (7) | 22 (22) | 27 (28) | 17 (17)
Pyrexia (General disorders) | 7 (8) | 13 (14) | 6 (6) | 18 (19) | 15 (15) | 12 (12)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 10 (10) | 7 (7) | 17 (18)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 14 (15)
Nasopharyngitis (Infections and infestations) | 15 (15) | 7 (7) | 15 (15) | 18 (19) | 19 (19) | 18 (18)
Pneumonia (Infections and infestations) | 12 (13) | 5 (5) | 4 (4) | 8 (8) | 15 (15) | 11 (11)
Respiratory tract infection (Infections and infestations) | 13 (13) | 6 (6) | 4 (4) | 19 (19) | 29 (31) | 17 (18)
Rhinitis (Infections and infestations) | 12 (12) | 8 (8) | 14 (16) | 15 (16) | 16 (16) | 12 (13)
Skin bacterial infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 22 (25) | 15 (15) | 19 (19)

LIMITATIONS AND CAVEATS:
The observed placental malaria rate was lower than expected causing the study to be under powered. After review of a futility analysis, the Sponsor and DSMB recommended allowing the study to conclude as planned and not to increase the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less